CLINICAL TRIAL: NCT03883763
Title: Non-inferiority Study of Hyperbaric Novabupi® (Bupivacaine S75: R25) Compared to Hyperbaric Neocaine® (Bupivacaine S50: R50) in Spinal Anesthesia in Lower Limbs Vascular Surgery
Brief Title: Hyperbaric Novabupi® in Spinal Anesthesia in Lower Limbs Vascular Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRT090
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-07

CONDITIONS: Spinal Anesthesia; Vascular Surgery
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Novabupi® 0.5% (bupivacaine S75:R25 + 8% glucose) (Experimental)
  Interventions: Drug: bupivacaine S75:R25 plus 8% glucose
- Hyperbaric Neocaine® 0.5% (bupivacaine S50:R50 + 8% glucose) (Active Comparator)
  Interventions: Drug: bupivacaine S50:R50 plus 8% glucose

INTERVENTIONS:
Drug: bupivacaine S75:R25 plus 8% glucose — Spinal anesthesia, 20 mg
  Arms: Hyperbaric Novabupi® 0.5% (bupivacaine S75:R25 + 8% glucose)
Drug: bupivacaine S50:R50 plus 8% glucose — Spinal anesthesia, 20 mg
  Arms: Hyperbaric Neocaine® 0.5% (bupivacaine S50:R50 + 8% glucose)

SUMMARY:
This is a multicenter, randomized, double-blind, active-controlled study to evaluate the non-inferiority of hyperbaric Novabupi® versus hyperbaric Neocaine® in spinal anesthesia in lower limbs vascular surgery.

The schedule consists of four visits: screening (visit 1); pre-anesthetic evaluation and randomization (visit 2); treatment (visit 3) and discharge from study (visit 4).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Both sexes
* Age between 18 and 80 years, inclusive
* ASA category I or II
* Indication of spinal anesthesia for varicose vein surgery in lower limbs with a maximum duration of 3 hours.

Exclusion Criteria:

* Contraindications to spinal anesthesia
* Hypersensitivity or intolerance to local anesthetics or to the components of formula
* Use of any anticoagulant, regardless of type until 60 days before entering the study
* Spinal cord injuries, peripheral neuropathies or any other neurological conditions leading to sensory and / or motor disorders
* Dementia, mental retardation and other major cognitive changes
* Obesity with body mass index (BMI) > 30 or difficulty in performing the puncture
* Anatomical difficulty in the spine in the opinion of the Investigator that can make puncture difficult
* Any previous surgical intervention of the spine
* Tattoo at the puncture site
* Participants with a history of alcohol or illicit drug abuse, as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th edition
* Pernicious anemia
* History of severe anaphylactic reactions or Steven-Johnson disease
* Changes in safety exams (applicable at the time of randomization):

  * International Normalized Ratio ≥ 1.4
  * Hemoglobin < 10 g / dL
  * Platelet count <100,000 / mm3
  * Glycemia> 200 mg / dL
  * Bradyarrhythmias: heart block with clinical repercussion in the investigator's opinion
  * Maximum of eight ventricular extrasystoles per minute, evident on the ECG
* Pregnancy or lactation
* Any other condition that, in the opinion of the Investigator, may lead to an increased risk for the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between arms from latency to T10 dermatome sensitive block | 20 minutes
  Time elapsed between the withdrawal of the needle at the end of the injection of the local anesthetic and the absence of response to sensorial stimuli in the region corresponding to the T10 dermatome
Comparison between arms from the duration of the sensory block | 24 hours
  Time elapsed between the withdrawal of the needle at the end of the local anesthetic injection and the presence of positive sensitivity by needle stimulation in the L5 dermatome

SECONDARY OUTCOMES:
Comparison between arms from the degree of motor blockage when blocking T10 sensitive | 20 minutes
  The motor block will be evaluated by the modified Bromage scale. The degree of motor block will be assessed when the sensory block reaches T10.
  The motor block will be evaluated every 5 minutes from the end of the anesthetic injection (time 0) through the modified Bromage scale:
  * 0 = without motor block,
  * 1 = blocked hip,
  * 2 = blocked hip and knee,
  * 3 = blocked hip, knee and ankle.
  Will be recorded:
  * the degree of motor blockage when the sensory block reaches T10,
  * the time to reach the maximum block,
  * time for full recovery (Bromage score 0).
Comparison between arms from the duration of the motor block | 24 hours
  Duration of motor block will be considered as the time interval between needle withdrawal after puncture and return to score 0 on the modified Bromage scale. Time will be recorded to reach grade 3 motor block and at the end of surgery. During anesthesia recovery, evaluations will be performed every 15 minutes
Comparison between arms from the highest level of sensory block | 3 hours
Comparison between arms from the time to reach the highest level of sensory block | 1 hour
Comparison between arms from the time for the 4-segment regression of the sensory block | 3 hours
  The height of the sensitive block will be evaluated every 5 minutes until the maximum level is reached. From this point, the height of the block will be evaluated every 10 minutes until the regression of 4 levels
Comparison between arms of respiratory and cardiovascular safety | 12 hours
  Evidenced by the incidence, severity and causality of clinically significant SpO2 changes.
  Every 5 minutes SpO2 will be recorded until completing 60 minutes, every 10 minutes until completing 120 minutes, every 20 minutes until 12 hours.
Comparison between arms of cardiovascular safety | 24 hours
  Evidenced by the incidence, severity and causality of clinically significant changes in blood pressure measured automatically by cardiac monitoring.
  Every 5 minutes blood pressure will be recorded until completing 60 minutes, every 10 minutes until completing 120 minutes, every 20 minutes until completing 180 minutes and every 30 minutes until complete recovery of the motor function.
Comparison between arms of cardiovascular safety | 12 hours
  Evidenced by the incidence, severity and causality of clinically significant changes in heart rate measured automatically by cardiac monitoring.
  Every 5 minutes heart rate will be recorded until completing 60 minutes, every 10 minutes until completing 120 minutes, every 20 minutes until completing 180 minutes and every 30 minutes until complete recovery of the motor function
Comparison between arms from the percentage of motor and sensory block failure | 20 minutes
  After the needle has been withdrawn, the anesthetic should be installed for up to 20 minutes. If no sensory and / or motor blockage is observed after this period, the Investigator will indicate that there was an anesthetic failure that should be classified as:
  A. total block failure (absence of anesthesia in sensory and motor aspects with preserved sensitivity of the perineal region) B. partial failure (when any area below the T10 dermatome shows signs of analgesia or motor block, but surgery can not be performed, requiring intense sedation or general anesthesia).
  In case of failure, the participant will be immediately discontinued from the study and the surgery will normally proceed with anesthetic procedure at the discretion of the Investigator. Anesthesia failure should be reported as an adverse event.
Comparison between arms from the occurrence of adverse events | 7 days
  Adverse event information will be collected from all participants on all visits

CONTACTS AND LOCATIONS:
Overall Officials: João B Garcia, MD/PhD, Principal Investigator — HUUFMA - Hospital Universitário da Universidade Federal do Maranhão
Locations (1):
- CEPEC, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No